CLINICAL TRIAL: NCT03148600
Title: Behavioural Treatment Following Ileo-Anal Pouch Formation:
Brief Title: Rehabilitation After Ileo-anal Pouch Surgery
Acronym: RAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St Vincent's Hospital Melbourne (Other)
Responsible Party: Principal Investigator, Angela Khera, Senior Clinician Physiotherapist, St Vincent's Hospital Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREC/16/SVHM/214
Record Dates: First submitted 2017-04-20; First posted 2017-05-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Colonic Pouches; Physical Therapy Modalities; Biofeedback
Keywords: Ileoanal pouch, pelvic floor exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Active Comparator): Pelvic floor and bowel behavioural training programme provided by physiotherapists over 2- 6 sessions within the 6 months following ileostomy closure for patients with an ileo-anal pouch
  Interventions: Behavioral: Pelvic floor and bowel behavioural training
- Standard arm (Placebo Comparator): Standard post-operative nursing and medical care provided in hospital clinic
  Interventions: Other: Standard arm

INTERVENTIONS:
Behavioral: Pelvic floor and bowel behavioural training — Physiotherapist-led pelvic floor muscle and bowel behavioural training
  Arms: Intervention arm
Other: Standard arm — Standard medical and nursing care
  Arms: Standard arm

SUMMARY:
Multi-centre, assessor-blinded, randomised controlled trial comparing physiotherapist-led behavioural intervention (including pelvic floor muscle training) to standard care, in the management of post-operative ileo-anal pouch patients.

ELIGIBILITY:
Inclusion Criteria:

* Proven (documented) history of Ulcerative Colitis or Familial Adenomatous Polyposis
* Proctocolectomy and awaiting ileo-anal pouch formation or have had ileo-anal pouch created and are waiting for stoma reversal or have had stoma reversal within the last 60 days

Exclusion Criteria:

* Primary sclerosing cholangitis
* Significant medical or psychiatric comorbidity that in the opinion of the investigators would interfere with bowel function or adherence to the protocol
* Clinically significant narcotic or substance abuse that in the opinion of the investigators would interfere with bowel function or adherence to the protocol
* Recognised eating disorder
* Non- English speaking or illiterate
* Pregnancy
* Current participant in another trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Colo Rectal Functional Outcome Score (COREFO) | 6 and 12 months following ileostomy reversal
  Between group comparison of outcome score - total and each of 5 domains

SECONDARY OUTCOMES:
Pouch Dysfunction score | 1,3,6 and 12 months following ileostomy closure
  Comparison of scores between groups
Quality of Life Short-Form 36 (SF-36) | Baseline, 3,6 and 12 months following ileostomy closure
  Quality of life SF-36 compared between groups - mental health domain, physical health domain and total score
Quality of Life EQ-5D | Baseline,3,6 and 12 months following ileostomy closure
  Scores from the EQ-5D will be compared between groups and quality adjusted life years (QALY) will be derived from EQ-5D.
Inflammatory Bowel Disease Questionnaire (IBDQ) | Baseline,3,6 and 12 months following ileostomy closure
  Disease specific quality of life score comparing groups
Hospital Anxiety and Depression Scale (HADs) | Baseline,3,6 and 12 months following ileostomy closure
  Psychological well being scores for anxiety and depression comparing groups
Brief Illness Perception Questionnaire | Baseline,3,6 and 12 months following ileostomy closure
  Between group comparison of cognitive and emotional perceptions of illness
Brief Cope | Baseline,3,6 and 12 months following ileostomy closure
  Between group comparison of coping styles and ability to cope with stress
New General Self-Efficacy Scale | Baseline,3,6 and 12 months following ileostomy closure
  Between group comparison of confidence in ability to perform tasks and achieve goals

OTHER OUTCOMES:
Patient Global Impression of Improvement and Satisfaction | 3,6 and 12 months following ileostomy closure
  Between group comparison of patient rating of improvement and satisfaction on 7-point Likert Scales
Adherence | 1,2,3,4,5 and 6 months following ileostomy closure
  Patient rating of their level of adherence to the training programme
Pelvic floor muscle function | Baseline and 6 months following ileostomy closure
  Transperineal measurements of displacement of puborectalis and change in anorectal angle with pelvic floor muscle contraction and with simulated defaecation
Cost to the healthcare system | Baseline, 6 and 12 months following ileostomy closure
  Compare health care utilisation between groups

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Kamm, MBBS,PhD, Principal Investigator — St Vincent's Hospital Melbourne
Locations (2):
- Australia (2):
  - St Vincent's Hospital, Fitzroy, Victoria
  - Alfred Health, Prahran, Victoria

IPD SHARING:
Plan to Share IPD: No